CLINICAL TRIAL: NCT05239403
Title: Delineating Gut Microbiome and Dietary Determinants Associated With Favorable Vaccine Response
Brief Title: Association Between Gut Microbiome and Dietary Determinants and Vaccine Response
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2020-1054; NCI-2021-09308 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-1054 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2022-02-03; First posted 2022-02-14 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (questionnaire, biospecimen collection): Participants complete questionnaires over 10-15 minutes up to 4 weeks prior to day of vaccination and undergo collection of blood samples up to 4 weeks before or on the day of vaccination and within 3 weeks post vaccination. Patients may also undergo collection of stool samples up to 4 weeks prior to day of vaccination.
  Interventions: Procedure: Biospecimen Collection; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood and stool samples
  Other Names: Biological Sample Collection; Biospecimen Collected
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This study evaluates the association between gut microbiome and dietary determinants and vaccine response. This study aims to learn if diet and the microbes (such as bacteria and viruses) found in your gut affect the body's immune response to the influenza vaccine.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the association of gut microbiome diversity with response to influenza vaccination as measured by vaccine-specific immune response.

SECONDARY OBJECTIVE:

I. To determine the gut microbial signatures and dietary patterns associated with response to influenza vaccination as measured by vaccine-specific post vaccine serum titers.

EXPLORATORY OBJECTIVES:

I. Interrogation of the overlap between the identified signature and excellent or poor responses to cancer immunotherapy (from our own published work and internal cohorts).

II. Identify components and determinants of the gut microbiome that could be modulated to enhance vaccine response.

OUTLINE:

Participants complete questionnaires over 10-15 minutes up to 4 weeks prior to day of vaccination and undergo collection of blood samples up to 4 weeks before or on the day of vaccination and within 3 weeks post vaccination. Patients may also undergo collection of stool samples up to 4 weeks prior to day of vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. MD Anderson employees and student employees with existing MRN
2. Must be able to donate blood
3. Participants must be age 18 or older
4. Participants must receive the seasonal influenza vaccine at MD Anderson through Employee Health
5. Participants must consent to gut microbiome profiling, REDCap-based dietary screening questionnaire (Appendix A) and survey (Appendix B), and vaccine immune response testing which requires one stool sample, and two blood draws

Exclusion Criteria:

1. Participants with a contraindication to the recommended annual influenza vaccine

Pregnant women may be included in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: MD Anderson employees
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-08-24 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Correlation between fecal microbiome diversity and seroconversion following influenza vaccination | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Wargo, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org